CLINICAL TRIAL: NCT00915057
Title: An Open Study to Investigate the Effects of Chronic Viral Hepatitis B or C on the Pharmacokinetics of Cholyl-lysyl-fluorescein (NRL972) Before, During and After Standard Treatment.
Brief Title: Effect of Chronic Viral Hepatitis on the Pharmacokinetics of NRL972.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Vice President Clinical Development, Norgine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NRL972-09/2008 (CHBC)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Hepatitis, Viral, Human
MeSH Terms: conditions — Hepatitis, Viral, Human | interventions — NRL972

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NRL972 (Experimental): Single 2mg intravenous dose of NRL972, administered on up to seven occasions
  Interventions: Drug: NRL972

INTERVENTIONS:
Drug: NRL972 — Single dose of NRL972 administered at baseline, at 3-monthly intervals during treatment for up to 12 months (or the end of treatment) and at 3 and 6 months after the end of treatment.

SUMMARY:
Little is known about the nature and extent of the disturbance in hepatic function and biliary hepatic clearance in chronic viral hepatitis, while the course of this disease, the functional implications and response to treatment are difficult to predict. This study aims to assess this in patients with chronic viral hepatitis B (CHB) and chronic viral hepatitis C (CHC) who are eligible for treatment in accordance with the established consensus guidelines in the involved countries. The pharmacokinetics of NRL972 will be determined at baseline (within one month of starting treatment), at 3-monthly intervals during treatment, for up to 12 months (or at the end of treatment), and at 3 and 6 months after the end on treatment. This will provide a clearer understanding regarding the use of the pharmacokinetics of NRL972 in detecting changes in biliary clearance during and after treatment for CHB and CHC.

ELIGIBILITY:
Inclusion Criteria:

Chronic viral hepatitis B

* Adult, male or female, age ≥ 18 years and < 65 years
* Body weight (BW) : 45 - 110 kg
* Body mass index (BMI) : 18 - 30 kg.m-2
* HBV Serology: HBsAg+ for ≥ 6 months (at the time of application for treatment)
* Serum ALT ≥ 1.5 times ULN ≥ 6 months (at the time of application for treatment)
* Positive liver biopsy within 24 months before screening visit
* Positive biopsy with signs of active disease (any level of activity by Knodell, METAVIR or ISHAK)
* HBV DNA counts determined by quantitative PCR: ≥ 20,000 IU/mL ALT < 10 times ULN
* HIV-Ab negative
* Non-cirrhotic liver disease (on histology within 24 months before screening visit)
* Not having been treated for chronic viral hepatitis previously ("de novo" i.e. "naïve")
* Eligible for treatment of chronic viral hepatitis in accordance with the national consensus guidelines pertinent to the country and site of conduct of the trial
* Willing and able to provide informed consent

Chronic viral hepatitis C

* Adult, male or female, age ≥ 18 years and < 65 years
* Body weight (BW) : 45 - 110 kg
* Body mass index (BMI) : 18 - 30 kg.m-2
* HCV-Ab+ for ≥ 6 months (at the time of application for treatment)
* HCV RNA counts > 10,000 U/L by quantitative PCR assay within the last 6 months (at the time of application for treatment)
* Positive liver biopsy within 24 months before application for treatment
* Positive biopsy with signs of fibrotic disease (levels of fibrosis METAVIR ≥ F1 or ISHAK ≥ F2)
* ALT < 10 times ULN
* HIV-Ab negative
* Non-cirrhotic liver disease (on histology within 24 months before screening visit)
* Not having been treated for chronic viral hepatitis previously ("de novo" i.e. "naïve")
* Eligible for treatment of chronic viral hepatitis in accordance with the national consensus guidelines pertinent to the country and site of conduct of the trial
* Willing and able to provide informed consent

Chronic viral hepatitis C plus chronic viral hepatitis B

* Patients with combined CHB and CHC will be managed (in terms of eligibility and standard treatment in accordance with the hepatitis type with predominant viral replication.

Exclusion Criteria:

Trial specific criteria: CHB, CHC & CHB+CHC

* Previous participation in the trial
* Participation in any other clinical trial within 30 days of entry to this protocol
* Treatment with any investigational drug within 30 days of entry to this protocol
* Non-response to previous treatment for chronic viral hepatitis
* Relapse after previous treatment for chronic viral hepatitis
* Any other known cause of liver disease other than chronic viral hepatitis B and/or C, including but not limited to hepatitis D, haemochromatosis, alpha1-antitrypsin deficiency, Wilson's disease, autoimmune hepatitis, drug-related liver disease
* Evidence of advanced liver disease, such as history or presence of ascites, bleeding varices, encephalopathy
* Patients with organ transplants
* Hypersensitivity to prospective standard treatment
* Any relevant co-morbidity, for instance, but not limited to:
* Limiting uncompensated psychiatric condition (e.g. severe depression, or a history of severe psychiatric disorder)
* CNS trauma or seizure disorder requiring medication
* Significant cardiovascular dysfunction within the past 6 months (e.g. angina, congestive cardiac failure, recent myocardial infarction, severe hypertension or significant arrhythmia)
* Patients with an ECG showing clinically significant abnormalities
* Poorly controlled diabetes mellitus
* Patients on haemodialysis
* Daily use of > 40 g alcohol
* Positive alcohol test at SCR-visit
* Evidence or suspicion of social drug abuse
* Positive drug test at SCR-visit
* Use of prohibited medication
* Suspicion or evidence that the subject is not trustworthy and reliable
* Suspicion or evidence that the subject is not able to make a free consent or to under-stand the information in this regard

Criteria specifically related to the standard treatment of chronic viral hepatitis

* Relevant clinical laboratory test abnormalities, for instance, but not limited to:

Haemoglobin (Hgb) <11 g dL-1 for women and <13 g dL-1 for men

White Blood Cell count (WBC) < 3,000 10 exp9/mL

Granulocyte count < 1,500 10 exp9/mL

Lymphocyte count < 500 10 exp9/mL

Platelets < 75,000 10 exp9/mL

Prothrombin time - INR > 1.4

Bilirubin > 25 micromol/L (except in functional hyperbilirubinaemia)

Albumin < 35 g/L

Serum creatinine > 133 micromol/L

Fasting blood glucose > 7.4 mmol/L for non-diabetic patients

HbA1c > 7% for diabetic patients

Positive auto-immune antibodies

TSH outside the normal range (for patients intended for interferon)

* Relevant co-morbidity, for instance, but not limited to:

Limiting uncompensated chronic pulmonary disease (e.g. chronic obstructive pulmonary disease)

Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids

Gout - (for patients intended for interferon)

Immunologically mediated disease (e.g. inflammatory bowel disease, Crohn's disease, ulcerative colitis, rheumatoid arthritis, idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune haemolytic anaemia, scleroderma, severe psoriasis, cryoglobulinaemia with vasculitis) - (for patients intended for interferon)

Patients with clinically significant retinal abnormalities - (for patients intended for interferon)

All females

* Positive pregnancy test
* Lactating
* Not using medically appropriate contraception and/or not willing to maintain such contraception during the treatment of chronic viral hepatitis and up to 6 months thereafter

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of NRL972 | Up to one hour post-dosing

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Gruss, MD, Study Director — Norgine
Locations (4):
- MHAT Sveti Ivan Rilski EAD, Sofia, Bulgaria
- Romania (3):
  - Clinical Institute Fundeni, Bucharest
  - Emergency Country Hospital Cluj, Cluj-Napoca
  - Private Clinic Algomed SRL, Timișoara